CLINICAL TRIAL: NCT01012193
Title: CYP 2C19 Polymorphism and Response to Adjunctive Cilostazol and High Maintenance-dose Clopidogrel in Patients Undergoing Elective Percutaneous Coronary Intervention
Brief Title: Adjunctive Cilostazol Versus High Maintenance-dose Clopidogrel According to Cytochrome 2C19 Polymorphism
Acronym: ACCEL-2C19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gyeongsang National University Hospital (Other)
Responsible Party: Young-Hoon Jeong/Assisstant professor, Gyeongsang National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GNUHIRB-2009-24
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: adjunctive cilostazol; high-MD clopidogrel; CYP 2C19 polymorphism; high risk patients
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cilostazol; BID protein, human; Clopidogrel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- adjunctive cilostazol (Active Comparator): adjunctive cilostazol 100mg bid to dual antiplatelet therapy
  Interventions: Drug: cilostazol 100mg bid or clopidogrel 150-mg daily
- high maintenance-dose clopidogrel (Active Comparator): double dose of clopidogrel 150mg/day
  Interventions: Drug: cilostazol 100mg bid or clopidogrel 150-mg daily

INTERVENTIONS:
Drug: cilostazol 100mg bid or clopidogrel 150-mg daily — Adjunctive cilostazol: cilostazol 100-mg bid +clopidogrel 75mg daily+aspirin 200mg daily High-MD clopidogrel: clopidogrel 150mg daly +aspirin 200mg daily

SUMMARY:
The purpose of this study is to determine the impact of adjunctive cilostazol versus high maintenance-dose clopidogrel on platelet inhibition in carriers and non-carriers of the loss-of-function CYP2C19 mutant allele.

DETAILED DESCRIPTION:
The additional platelet inhibition with clopidogrel, a thienopyridine inhibitor of the platelet P2Y12 adenosine diphosphate (ADP) receptor, has reduced the risk of ischemic events after coronary stent implantation. Because of inter-individual variability in platelet response to clopidogrel, a significant proportion of suboptimal platelet inhibition has been reported. In addition, persistent residual platelet reactivity measured with platelet function testing has shown the association with the cardiovascular outcomes after percutaneous coronary intervention (PCI).

Various clinical factors and genetic polymorphisms have been studied to predict the degree of antiplatelet response to clopidogrel. Interestingly, recent studies found that carriers of the loss-of-function hepatic cytochrome (CYP) 2C19 allele had significantly lower levels of the active metabolite of clopidogrel, diminished platelet inhibition, and a higher rate of major adverse cardiovascular events than did non-carriers, in the setting of PCI and acute coronary syndrome (ACS). These findings raise the need of solutions to overcome enhanced post-clopidogrel platelet reactivity by the influence of the loss-of-function CYP2C19 allele. Increasing the dose of clopidogrel and new potent P2Y12 antagonists (such as prasugrel) may be alternative antiplatelet regimens in patients with the loss-of-function CYP variant.

Cilostazol reversibly induces platelet inhibition via its blockade of phosphodiesterase (PDE) type 3 and is catalysed mainly by CYP3A. A recent study demonstrated that adjunctive cilostazol to dual antiplatelet therapy (triple antiplatelet therapy) intensified platelet inhibition as compared with a high maintenance-dose (MD) of 150 mg/day. Therefore, triple antiplatelet therapy could also be an alternative antiplatelet therapy to improve platelet inhibition and clinical outcomes in carriers of CYP2C19 mutant allele.

We compared the enhanced inhibition of platelet aggregation by adjunctive cilostazol 100 mg twice daily versus high-MD clopidogrel 150 mg/day in patients treated with elective coronary stenting, according to the CYP2C19 polymorphism.

ELIGIBILITY:
Inclusion Criteria:

* Significant coronary artery stenosis (>70% by visual estimate)
* Elective coronary stent implantation

Exclusion Criteria:

* Acute myocardial infarction
* Active bleeding and bleeding diatheses
* Hemodynamic instability
* Oral anticoagulation therapy with warfarin
* Use of peri-procedural glycoprotein IIb/IIIa inhibitors
* Contraindication to antiplatelet therapy
* Left ventricular ejection fraction < 30%
* Leukocyte count < 3,000/mm3, platelet count < 100,000/mm3, AST or ALT ≥ 3 times upper normal
* Serum creatinine level ≥ 3 mg/dL
* Stroke within 3 months
* Noncardiac disease with a life expectancy < 1 year
* Inability to follow the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Reduction of maximal platelet aggregation according to CYP 2C19 polymorphism | 30-day therapy

SECONDARY OUTCOMES:
Reduction of late platelet aggregation, reduction of P2Y12 reaction unit, and the rate of high post-clopidogrel platelet reactivity according to CYP 2C19 polymorphism | 30-day therapy

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoon Jeong, MD, PhD, Principal Investigator — Gyeongsang National University Hospital
Locations (1):
- Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do, South Korea

REFERENCES:
- [Derived] Jeong YH, Tantry US, Park Y, Kwon TJ, Park JR, Hwang SJ, Bliden KP, Koh EH, Kwak CH, Hwang JY, Kim S, Gurbel PA. Pharmacodynamic effect of cilostazol plus standard clopidogrel versus double-dose clopidogrel in patients with type 2 diabetes undergoing percutaneous coronary intervention. Diabetes Care. 2012 Nov;35(11):2194-7. doi: 10.2337/dc11-2351. Epub 2012 Jul 26. PMID 22837373
- [Derived] Kim IS, Jeong YH, Park Y, Yoon SE, Kwon TJ, Park JR, Hwang SJ, Koh EH, Kwak CH, Hwang JY, Kim S. Interaction analysis between genetic polymorphisms and pharmacodynamic effect in patients treated with adjunctive cilostazol to dual antiplatelet therapy: results of the ACCEL-TRIPLE (Accelerated Platelet Inhibition by Triple Antiplatelet Therapy According to Gene Polymorphism) study. Br J Clin Pharmacol. 2012 Apr;73(4):629-40. doi: 10.1111/j.1365-2125.2011.04131.x. PMID 22007612
- [Derived] Hwang SJ, Jeong YH, Kim IS, Park KS, Kang MK, Koh JS, Park JR, Park Y, Koh EH, Kwak CH, Hwang JY, Kim S. Cytochrome 2C19 polymorphism and response to adjunctive cilostazol versus high maintenance-dose clopidogrel in patients undergoing percutaneous coronary intervention. Circ Cardiovasc Interv. 2010 Oct;3(5):450-9. doi: 10.1161/CIRCINTERVENTIONS.110.949859. Epub 2010 Sep 7. PMID 20823393
- See also: Pubmed release of ACCEL study — http://www.ncbi.nlm.nih.gov/pubmed/20823393